CLINICAL TRIAL: NCT03590977
Title: Evaluation the Efficacy of a Herbal Licorice on Reducing Salivary Streptococcus Mutans Levels (A Randomized Clinical Trial)
Brief Title: Efficacy of Licorice on Reducing Salivary Streptococcus Mutans Versus Chlorohexidine in Caries Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nancy Helmy Blamon Mikhael, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-07-5
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Caries, Dental
Keywords: Streptococcus Mutans; licorice; chlorohexidine; caries index
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- licorice extract mouthwash (Experimental): administration of a mouthwash containing licorice as a preventive measure to high caries risk patients (faculty of pharmacy, cairo university)
  Interventions: Other: licorice extract mouthwash
- chlorohexidine mouthwash (Placebo Comparator): administration of chlorohexidine 0.2% in 1:1 diluation mouthwash that is broad spectrum antimicrobial activity to high caries risk patients
  Interventions: Other: chlorohexidine mouthwash

INTERVENTIONS:
Other: licorice extract mouthwash — mouth rinse that contains a natural herbal licorice root extract used as a preventive measure that reduce caries index.
  Arms: licorice extract mouthwash
Other: chlorohexidine mouthwash — mouth wash that contains chlorohexidine as an active component
  Arms: chlorohexidine mouthwash

SUMMARY:
To compare the effect of a natural herbal licorice containing preventive measure alternative to chlorohexidine preventive measure to decrease the effect of streptococcus mutans.

DETAILED DESCRIPTION:
A total number of fifty-two patients will be enrolled in the study. They will be divided into two groups: study group and control group. Study group will be subjected to licorice mouthwash and the control will be subjected to chlorohexidine mouth wash. Salivary bacterial count will be evaluated for both groups.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* co-operative patients
* not allergic to licorice
* not allergic to chlorohexidine

Exclusion Criteria:

* pregnancy
* allergic patients to licorice
* allergic patients to chlorohexidine
* lack of compliance
* evidence of parafunctional habits
* patients with periodontal disease
* xerostomia
* participants that receive any microbial agent two weeks prior to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
salivary bacterial count | after one week
  streotococcus mutans bacterial count

CONTACTS AND LOCATIONS:
Overall Officials: nancy helmy, Msc, Principal Investigator — Faculty of Dentistry, Cairo univerisity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almaz ME, Sonmez IS, Okte Z, Oba AA. Efficacy of a sugar-free herbal lollipop for reducing salivary Streptococcus mutans levels: a randomized controlled trial. Clin Oral Investig. 2017 Apr;21(3):839-845. doi: 10.1007/s00784-016-1827-y. Epub 2016 Apr 30. PMID 27129589
- [Background] Jain E, Pandey RK, Khanna R. Liquorice root extracts as potent cariostatic agents in pediatric practice. J Indian Soc Pedod Prev Dent. 2013 Jul-Sep;31(3):146-52. doi: 10.4103/0970-4388.117964. PMID 24021323